CLINICAL TRIAL: NCT02899286
Title: A Phase II Open-label Study of the Efficacy and Safety of Recombinant Human Arginase 1 (PEG-BCT-100) in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Efficacy and Safety Study of Recombinant Human Arginase 1 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bio-Cancer Treatment International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCT-100-007
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; AML; pegylated recombinant human arginase; PEG-BCT-100
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BCT-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-BCT-100 (Experimental): PEG-BCT-100 (PEGylated recombinant human arginase)
  Interventions: Biological: PEG-BCT-100

INTERVENTIONS:
Biological: PEG-BCT-100 — PEGylated recombinant human arginase

SUMMARY:
To evaluate the efficacy of PEG-BCT-100 in patients with relapsed or refractory acute myeloid leukemia (AML) in terms of remission rate.

DETAILED DESCRIPTION:
This is a phase 2, non-randomised, open-label study that aims at evaluating the efficacy of single agent PEG-BCT-100 in adult patients with relapsed/refractory AML. Eligible patients will receive intravenous (IV) infusion of PEG-BCT-100 weekly until disease progression, unacceptable drug-related toxicity(ies), allogeneic haematopoietic stem cell transplantation or withdrawal of subject consent.

Pharmacokinetic (PK) of PEG-BCT-100 and pharmacodynamics (PD) activity of PEG-BCT-100 on arginine depletion will be evaluated throughout the study. Plasma arginine level, intracellular blast arginine level (IBAL) in peripheral blood (PB) and bone marrow (BM) will be measured at specific time points. PEG-BCT-100 will be given once weekly at 1600 Units/kg (2.7mg/kg) per dose for three weeks (Cycle 1). If the post-treatment IBAL-BM examined within 5 days prior to each cycle fails to drop at least 70% from baseline value and disease response fails to achieve complete remission (CR) or complete remission with incomplete blood count recovery (CRi), PEG-BCT-100 may be increased to 2500 U/kg (the maximum tolerated dose as reported previously) at investigator's discretion. Disease response will be assessed within 5 days prior to each cycle according to the International Working Group (IWG) AML Response Criteria.

Safety and toxicity will be assessed through physical examinations, vital signs, blood tests and urinalysis throughout the study. Adverse event (AE) and serious adverse events (SAE) will be reported according to the National Cancer Institute Common Toxicity Criteria for Adverse Events version 4.03 (CTCAE v4.03) until 28 days after the last dose of PEG-BCT-100.

Immunogenicity response including anti-drug antibody (ADA) level and neutralizing antibody level will be assessed weekly for the first 2 cycles of PEG-BCT-100, pre-dose of each cycle thereafter and End of Study (EoS). Specific response predictive biomarkers in circulating and BM blasts, and emerging genetic markers will also be explored in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥18 year-old at the time of informed consent
2. Documented relapsed or refractory AML after at least two standard chemotherapy regimen or in whom the treating physicians considered unfit for further chemotherapy treatment
3. The Eastern Cooperative Oncology Group (ECOG) performance status equal or less than 2
4. Patients from whom valid consent is obtained

Exclusion Criteria:

1. Patients who have received any induction chemotherapy, investigational treatment and arginine depleting agent within 2 weeks prior to the start of the PEG-BCT-100 (not including hydroxyurea or thioguanine)
2. Any toxic effects (except hair loss) of the prior therapy have not been resolved to Grade 1 or less according to National Cancer Institute Common Terminology Criteria for Adverse Events
3. Total bilirubin > 1.5 x Upper Limit of Normal (ULN) not related to haemolysis or Gilbert's disease, and ratio of concentrations of aspartate transaminase and alanine transaminase (AST/ALT) > 5 x ULN
4. Creatinine > 2 x ULN or estimated glomerular filtration rate using Modification of Diet in Renal Disease formula < 60 ml/min/1.73 m2
5. Second active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
6. Uncontrolled concomitant illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia
7. History of HIV-1 seropositivity
8. Active infection not adequately responding to appropriate therapy
9. Patient is pregnant or lactating
10. Female with childbearing potential who is not willing to use contraceptive methods which, in the opinion of the investigator, are effective and adequate while on study treatment and for 6 months after the last dose of study treatment
11. Male with a female partner with childbearing potential who is not willing to use contraceptive methods which, in the opinion of the investigator, are effective and adequate while on study treatment and for 6 months after the last dose of study treatment
12. Any condition that is unstable or can jeopardize the safety of the patients and their compliance to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | 3 years

SECONDARY OUTCOMES:
Overall response rate (ORR) | 3 years
  proportion of patients achieving CR or CRi or partial remission (PR)
Duration of remission | 3 years
Time to progression (TTP) | 3 years
Progression-free survival (PFS) | 3 years
Overall survival (OS) | 3 years
AE and SAE | 3 years
  Incidence of AE and SAE by severity grading as assessed according to CTCAE v4.03
PK - Area under the plasma concentration versus time curve (AUC) | 2 years
PK - Peak plasma concentration of PEG-BCT-100 after administration (Cmax) | 2 years
PK - Lowest concentration that PEG-BCT-100 reaches before the next dose is administered (Cmin) | 2 years
PK - clearance | 2 years
PK - volume of distribution | 2 years
PK - elimination half-life | 2 years
PD | 2 years
  arginine depletion
PK/PD relationship | 2 years
  dose response
Anti-drug antibody (ADA) | 2 years
  amount of ADA in patient sample (ng/mL)
neutralizing anti-drug antibody (nADA) | 2 years
  amount of nADA in patient sample (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Anskar Leung, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided